CLINICAL TRIAL: NCT02029820
Title: RenalGuard System for Prevention of Contrast Induced Nephropathy - A Randomized Trial
Brief Title: RenalGuard System for Prevention of Contrast Induced Nephropathy
Acronym: REPRECIN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sao Lucas da PUCRS (Other)
Responsible Party: Principal Investigator, Vitor Osorio Gomes, MD, PhD, Hospital Sao Lucas da PUCRS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11/05339
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Radiographic Contrast Agent Nephropathy
Keywords: Contrast Nephropathy; Prevention; Renalguard

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RenalGuard (Active Comparator): Hydration with the device renalguard
  Interventions: Device: RenalGuard
- Saline (No Intervention): Hydration with saline 1ml/Kg/h for 12h

INTERVENTIONS:
Device: RenalGuard — Intravenous saline hydration matched with urine output, using the device Renalguard
  Arms: RenalGuard

SUMMARY:
The purpose of this study is to determine whether hydration with intravenous saline matched with urine output, using the device RenalGuard is superior to standard hydration with saline to prevent contrast-induced nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* serum creatinine >1.2mg/dl
* glomerular filtration rate (GFR) < 60ml/min

Exclusion Criteria:

* acute renal failure
* use of radiological contrast in the latest 7 days
* Current use of N-acetylcysteine or hydration of sodium bicarbonate
* Patients in dialysis
* Emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of contrast-induced nephropathy | 72 hours
  Contrast-induced nephropathy defined as an increase of serum creatinine of 0.5mg/dl or 25% in pre procedure serum creatinine at 72h after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Vitor O Gomes, MD,PhD, Principal Investigator — Hospital Sao Lucas
Locations (1):
- Hospital São Lucas -PUCRS, Serviço de Hemodinâmica, Porto Alegre, Rio Grande do Sul, Brazil